CLINICAL TRIAL: NCT04442412
Title: Prephase Treatment With Prednisone +/- Vitamin D Supplementation Followed by Immunochemotherapy in Elderly Patients With Diffuse Large B-Cell Lymphoma (DLBCL) A Randomized, Open Label, Phase III Study by Fondazione Italiana Linfomi.
Brief Title: Prephase Treatment With Prednisone +/- Vitamin D Supplementation Followed by Immunochemotherapy
Acronym: FIL_PREVID
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: GRADE Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIL_PREVID
Record Dates: First submitted 2020-05-26; First posted 2020-06-22 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B-Cell Lymphoma; Elderly Patients
Keywords: Vitamin D; prednisone +/- Vitamin D supplementation; randomized, open label, phase III
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter, randomized phase III trial. The study plans to randomize patients with a 1 to 1 ratio to Arm A (Standard arm) or Arm B (Experimental arm). All patients of both arms will receive a prephase with oral prednisone before 6 cycles Q21 of immunochemotherapy with R-CHOP or R-miniCHOP at standard doses; patients in the Experimental arm (Arm B) will receive also a prephase therapy with VitD and a supplementation of VitD during the intere period of immunochemotherapy according to a prefixed schedule. Choice of type of immunochemotherapy will not rely on Comprehensive Geriatric Assessment result, but treatment at reduced doses with R-miniCHOP is highly recommended option for UNFIT and FRAIL patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm B (Experimental): (Experimental): Patients randomized to Arm B will receive a prephase with oral prednisone and a prephase therapy with VitD according to the below reported schedule followed by 6 courses of R-CHOP or R-miniCHOP every 21 days.
  Schedule for VitD supplementation: 25,000 U/day starting on day -6:
  daily loading dose for 7 days if 25 VitD baseline level 20-40 ng/ml daily loading dose for 14 days if 25 VitD baseline level < 20 ng/ml followed by weekly maintenance supplementation of 25,000 U for the entire duration of immunochemotherapy (6 courses every 21 days - 18 weeks), regardless of the baseline level of 25 VitD.
  Interventions: Drug: Vitamin D3 (Cholecalciferol); Drug: RCHOP o R-miniCHOP at standard doses
- Arm A (Standard arm) (Other): Patients randomized to Arm A will receive a prephase with oral prednisone followed by 6 courses of R-CHOP or R-miniCHOP every 21 days.
  If patients randomized to arm A are already on VitD, they are allowed to continue receiving VitD supplementation at a dose that can be considered part of the standard of care and does not exceed the maximum standard VitD dose recommended for general adult and elderly population , up to 10,000 U/week VitD
  Interventions: Drug: RCHOP o R-miniCHOP at standard doses

INTERVENTIONS:
Drug: Vitamin D3 (Cholecalciferol) — patients in the Experimental arm (Arm B) will receive also a prephase therapy with VitD and a supplementation of VitD during the intere period of immunochemotherapy according to a prefixed schedule. Choice of type of immunochemotherapy will not rely on Comprehensive Geriatric Assessment (CGA) result, but treatment at reduced doses with R-miniCHOP is highly recommended option for UNFIT and FRAIL patients.
  Arms: Arm B (Experimental):
Drug: RCHOP o R-miniCHOP at standard doses — Patients on both arms receive pre-treatment with prednisone oral before 6 cycles of 21 days each of immunochemotherapy with RCHOP
  o R-miniCHOP at standard doses

SUMMARY:
This is an open-label, multicenter, randomized phase III trial. The study plans to randomize patients with a 1 to 1 ratio to Arm A (Standard arm) or Arm B (Experimental arm).

All patients of both arms will receive a prephase with oral prednisone before 6 cycles Q21 of immunochemotherapy with R-CHOP or R-miniCHOP at standard doses; patients in the Experimental arm (Arm B) will receive also a prephase therapy with VitD and a supplementation of VitD during the intere period of immunochemotherapy according to a prefixed schedule. Choice of type of immunochemotherapy will not rely on Comprehensive Geriatric Assessment result, but treatment at reduced doses with R-miniCHOP is highly recommended option for UNFIT and FRAIL patients.

DETAILED DESCRIPTION:
After the patient signs the written informed consent the patient will enter the screening phase planning baseline assessments and will be randomly allocated with a 1 to 1 ratio to Arm A (Standard arm) or Arm B (Experimental arm).

Patients randomized to Arm A will receive a prephase with oral prednisone (50 mg for 7 days [day -6 to day 0]) followed by 6 courses of R-CHOP or R-miniCHOP every 21 days.

If patients randomized to arm A are already on VitD, they are allowed to continue receiving VitD supplementation at a dose that can be considered part of the standard of care and does not exceed the maximum standard VitD dose recommended for general adult and elderly population , up to 10,000 U/week VitD .

If clinically indicated at treating physician judgement, patients could receive 1 mg of vincristine on the first day of prephase ; in this case vincristine administration in cycle 1 of immunochemotherapy should be skipped, in patients receiving R-miniCHOP; reduced to 1 mg, in patients receiving R-CHOP.

Patients randomized to Arm B will receive a prephase with oral prednisone and a prephase therapy with VitD according to the below reported schedule followed by 6 courses of R-CHOP or R-miniCHOP every 21 days.

Schedule for VitD (Cholecalciferol) supplementation: 25,000 U/day starting on day -6:

daily loading dose for 7 days if 25 VitD baseline level 20-40 ng/ml daily loading dose for 14 days if 25 VitD baseline level < 20 ng/ml followed by weekly maintenance supplementation of 25,000 U for the entire duration of immunochemotherapy (6 courses every 21 days - 18 weeks), regardless of the baseline level of 25 VitD.

If clinically indicated at treating physician judgement, patients could receive 1 mg of vincristine on the first day of prephase (DAY -6); in this case vincristine administration in cycle 1 of immunochemotherapy should be: skipped, in patients receiving R-miniCHOP; reduced to 1 mg, in patients receiving R-CHOP.

Patients with 25(OH)VitD levels <30 ng/ml on d1 cycle 2 will receive and additional loading phase of Cholecalciferol 25,000 U/day for 7 days and then 25,000 U once weekly for the duration of immunochemotherapy.

Patients may continue with VitD supplementation after the end of the immunochemotherapy at a (reduced) standard dose of 25,000 U once a month for up to 2 years from end of immunochemotherapy.

Patients experimenting toxicity leading to a delay in treatment administration > 4 weeks will discontinue study treatment and will be addressed to a salvage treatment: these patients will be followed-up for survival until the end of the study.

Consolidation radiotherapy:

ELIGIBILITY:
Inclusion criteria

1. Histologically documented diagnosis of Diffuse Large B-cell Lymphoma or Follicular grade IIIb lymphoma, as defined in the 2017 edition of the World Health Organization (WHO) classification.
2. Age ≥ 65 years
3. Comprehensive Geriatric Assessment performed at baseline, before start of any treatment.
4. Eastern Cooperative Oncology Group performance status (PS) ≤3
5. Eligibility for anthracycline containing regimen (R-CHOP or R-miniCHOP)
6. No previous treatment for DLBCL or Follicular grade IIIb lymphoma
7. Ann Arbor stage I-IV
8. At least one site of measurable nodal disease at baseline ≥ 1.5 cm in the longest transverse diameter as determined by CT scan ; or one metabolic active site of disease at baseline FDG-PET scan
9. Serum basic levels of Vitamin D [25 (OH) VitD] ≤ 40 ng / ml;
10. Adequate hematological counts defined as follows:

    * Absolute Neutrophil count > 1.5 x 109/L unless due to bone marrow involvement by lymphoma
    * Platelet count ≥ 80.000/mm3 unless due to bone marrow involvement by lymphoma
11. Adequate renal function defined as follows:

    - Creatinine ≤ 2 mg/dL, unless secondary to lymphoma
12. Adequate hepatic function defined as follows:

    - Bilirubin ≤ 2 mg/dL unless secondary to lymphoma
13. LVEF > 50% at bidimensionally echocardiogram
14. Life expectancy ≥ 6 months
15. Subject understands and voluntarily signs an informed consent form approved by an Independent Ethics Committee , prior to the initiation of any screening or study-specific procedures
16. Subject must be able to adhere to the study visit schedule and other protocol requirements
17. Men must agree to use one of the below reported acceptable method of contraception for the duration of the study and for 3 months after receiving the last dose of immunochemotherapy, and to not donate sperm while on study.

Exclusion criteria

1. Histological diagnosis different from Diffuse large B-Cell Lymphoma or Follicular grade IIIb lymphoma, including diagnosis of HGBL, with rearrangement of MYC, BCL2 and/or BCL6 (double-hit)
2. Use of VitD supplementation as standard of care at dose higher than 10,000 U/week
3. Suspect or clinical evidence of CNS involvement by lymphoma
4. Contraindication to the use of rituximab
5. Contraindication to the use of VitD supplementation (Hypercalcemia/Hyperphosphatemia)
6. Subject has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, investigational therapy, including targeted small molecule agents within 14 days prior to the first dose of study drug
7. Significant history of neurologic, psychiatric, endocrinological, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent
8. Any history of other active malignancies within 2 years prior to study entry, with the exception of adequately treated in situ carcinoma of the cervix uterine, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin or limited stage surgically removed breast cancer or adequately treated with radiation therapy or limited stage prostate carcinoma surgically removed or adequately treated with radiation therapy or previous malignancy confined and surgically resected with curative intent
9. Evidence of other clinically significant uncontrolled condition including, but not limited to:

   * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
   * Chronic hepatitis B virus or hepatitis C requiring treatment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | at the end of treatment - 54 months
  Progression-Free Survival

SECONDARY OUTCOMES:
Overall Survival | at the end of treatment - 54 months
  Overall Survival
Event Free Survival | at the end of treatment - 54 months
  Event Free Survival (EFS)
Response rate | at the end of treatment - 54 months
  Response rate
Early death rate | at the end of treatment - 54 months
  Early death rate
Rate of ECOG changes after prephase | at the end of treatment - 54 months
  Rate of ECOG changes after prephase
Rate of patients who maintain 25(OH)VitD levels | At the beginning of Cycle 2 (each cycle is 21 days)
  Rate of patients who maintain 25(OH)VitD levels
Rate of 25(OH)VitD correction (VitD supplementation arm) | At the beginning of Cycle 2 (each cycle is 21 days)
  Rate of 25(OH)VitD correction (VitD supplementation arm)
time-to-deterioration physical functioning and fatigue | At the beginning of Cycle 2 (each cycle is 21 days)
  time-to-deterioration physical functioning and fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Merli, Dott., Principal Investigator — Reggio Emilia - Azienda Unitа Sanitaria Locale-IRCCS
Locations (49):
- Italy (49):
  - SC Ematologia Spedali Civili, Brescia, BS
  - UO Ematologia e CTMO di Piacenza, Piacenza, PC
  - Ospedale Oncologico regionale CROB, Rionero in Vulture, Piacenza
  - A.O. SS. Antonio e Biagio e Cesare Arrigo - S.C. Ematologia, Alessandria
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona, Ancona
  - Ascoli Piceno - Ospedale C.e G. Mazzoni - U.O.C. di Ematologia, Ascoli Piceno
  - Aviano - Centro Riferimento Oncologico - S.O.C. Oncologia Medica A, Aviano
  - Barletta - Ospedale "Monsignor Raffaele Dimiccoli" - Ematologia, Barletta
  - Bergamo - Cliniche Humanitas Gavazzeni - Oncologia - Cliniche Humanitas Gavazzeni, Bergamo
  - Biella - Ospedale Degli Infermi - S.C. Oncologia, Biella
  - Campobasso - Universitа Cattolica del Sacro Cuore - Ematologia, Campobasso
  - Castelfranco Veneto - Ospedale di Castelfranco Veneto - Ematologia, Castelfranco Veneto
  - Unità Funzionale di Ematologia AOU Careggi, Florence
  - Frosinone - Presidio Ospedaliero F. Spaziani - UOC Ematologia, Frosinone
  - Matera - Ospedale Madonna delle Grazie - Ematologia, Matera
  - Meldola - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) - Ematologia, Meldola
  - Mestre - Ospedale Dell Angelo - U.O. Ematologia, Mestre
  - SC Ematologia AO Niguarda Cà Granda, Milan
  - Monza - ASST MONZA Ospedale S. Gerardo - Ematologia, Monza
  - Napoli - AOU Universitа degli Studi della Campania Luigi Vanvitelli - Oncologia Medica ed Ematologia, Napoli
  - Università del Piemonte Orientale - Novara, Novara
  - Padova - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua
  - Pagani - Presidio ospedaliero "A. TORTORA" - U.O. Onco-ematologia, Pagani
  - Palermo - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - Palermo - AOU Policlinico Giaccone - Ematologia, Palermo
  - UO Ematologia Università - Policlinico San Matteo, Pavia
  - Pescara - P.O. Spirito Santo di Pescara - UOS Dipartimentale - Centro di diagnosi e Terapia dei linfomi, Pescara
  - Potenza - AOR San Carlo, Potenza
  - UO Ematologia Ospedale Santa Maria delle Croci, Ravenna
  - Reggio Emilia - AO Santa Maria Nuova, Reggio Emilia
  - UO Ematologia - Ospedale degli Infermi, Rimini
  - Roma - IRCCS Spallanzani - Servizio di Ematologia in malattie infettive, Roma
  - Roma - Ospedale S. Camillo - Ematologia, Roma
  - Roma - Policlinico Universitario Campus Bio-Medico - Ematologia - Trapianto cellule staminali - Medicina Trasfusionale e Terapia cellulare, Roma
  - Università Cattolica S. Cuore, Ematologia, Roma
  - Università La Sapienza Ematologia, Roma
  - UOC Ematologia - A.O. Sant'Andrea, Roma
  - Salerno - Ematologia e Trapianti A.O. San Giovanni di Dio e Ruggi D Aragona - U.O. Ematologia, Salerno
  - San Giovanni Rotondo - Casa Sollievo della Sofferenza - U.O. Ematologia, San Giovanni Rotondo
  - Sassari - AOU di Sassari - Ematologia, Sassari
  - UOC Medicina Interna MO DH Oncologico, Sassuolo
  - UOC Ematologia, AOU Senese, Siena
  - Univ. Perugia Sede Terni - Oncoematologia, Terni
  - AOU Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - SC. Ematologia A.O. Città della Salute e della Scienza, Torino
  - Torino - San Giovanni Bosco - ASL Cittа di Torino - SSD di Ematologia e Malattie Trombotiche, Torino
  - Trieste - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - SC Ematologia, Trieste
  - Udine - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) - SOC Clinica Ematologica, Udine
  - ULSS 8 Berica - Ospedale S. Bortolo - Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: No
This is an open-label, multicenter, randomized phase III trial. The study plans to randomize patients with a 1:1 ratio to Arm A (Standard arm) or Arm B (Experimental arm). All patients of both arms will receive a prephase with oral prednisone before 6 cycles Q21 of immunochemotherapy with R-CHOP or R-miniCHOP at standard doses; patients in the Experimental arm (Arm B) will receive also a prephase therapy with VitD and a supplementation of VitD during the intere period of immunochemotherapy according to a prefixed schedule. Choice of type of immunochemotherapy will not rely on Comprehensive Geriatric Assessment (CGA) result, but treatment at reduced doses with R-miniCHOP is highly recommended option for UNFIT and FRAIL patients.